CLINICAL TRIAL: NCT01749033
Title: A New Insertion Technique for Laryngeal Mask Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David Walega, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STU00046964
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Airway Morbidity
Keywords: Intubation; Airway; Laryngeal Mask Airway

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 classic (Active Comparator): Group 1 Using the classic inserting technique and completely deflated LMA (Laryngeal Mask Airway)recommended in the LMA manual.
  Interventions: Other: Group 1 Classic
- Group 2 pre inflated (Active Comparator): Group 2 (pre-inflated): Using the recommended inserting technique with the pre-inflated volume that exists in a LMA (Laryngeal Mask Airway) from the manufacturer
  Interventions: Other: Group 2 pre-inflated
- Group 3 ELL-PIC technique (Active Comparator): Group 3 (ELL-PIC): Using the ELL-PIC technique.
  Interventions: Other: Group 3 ELL-PIC

INTERVENTIONS:
Other: Group 1 Classic — Active Comparator: Group 1 classic
  Group 1 Using the classic inserting technique and completely deflated LMA recommended in the LMA manual.
  Arms: Group 1 classic
Other: Group 2 pre-inflated — Group 2 (pre-inflated): Using the recommended inserting technique with the pre-inflated volume that exists in a LMA (Laryngeal Mask Airway) from the manufacturer.
  Arms: Group 2 pre inflated
Other: Group 3 ELL-PIC — Group 3 (ELL-PIC): Using the ELL-PIC technique
  Arms: Group 3 ELL-PIC technique

SUMMARY:
A laryngeal mask airway ("LMA") is an airway device that is commonly used and placed under general anesthesia to facilitate ventilation of the patient's lungs while anesthetized. It is similar to an "endotracheal tube" (a breathing tube) but is less invasive. It is also placed as a backup when the Anesthesiologist is unable to pass a breathing tube and the patient is not adequately ventilating. Unfortunately, an LMA may lead to complications similar to those of breathing tube placement, such as sore throat and hoarse voice. Previous studies have examined several variables that may affect how often complications occur; these variables include giving anti-inflammatory medications and inflating the LMA to different pressures (the "working" end of the LMA, which rests in the patient's throat, has a cuff that is inflated to provide a seal). We are studying the effect of the PLACEMENT TECHNIQUE on postoperative sore throat, hoarse voice, and difficulty swallowing. We will be using 3 placement techniques - the traditional placement technique, a slightly different traditional placement technique, and a new technique, abbreviated the "ELLIA" method. The hypothesis of this study is that a new LMA insertion technique will have no difference in postoperative pharyngolaryngeal morbidity including sore throat, dysphagia and dysphonia.

DETAILED DESCRIPTION:
The LMA will be inserted based on one of three methods randomly assigned to each patient. The ELLIA technique involves gently lifting the patient's laryngeal structures (throat) while placing the LMA to oppose the force of gravity. Whereas the traditional method of placement involves guiding the LMA through the pharynx with a finger inserted into the pharynx, the ELLIA method avoids this step. General anesthesia will be maintained at the discretion of the Anesthesiologist throughout the surgical procedure. At the end of the case, as would normally occur, the LMA will be removed from the patient's airway and the patient will be taken to the PACU, where he or she will be cared for as usual. At one and two hours postoperatively, blinded research assistants will assess the patient for sore throat, hoarse voice, and difficulty swallowing. Finally, at 24 hours the patient will receive a telephone call from a blinded research assistant assessing for the same outcomes. These data will be collected and presented.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists patient fitness category) I, II, III
* Age 18-90
* General anesthetic for where LMA (Laryngeal Mask Airway) placement is not contraindicated will be included

Exclusion Criteria:

* Small mouth opening
* Preoperative sore throat/dysphagia/dysphonia
* Patients at increased risk for aspiration
* Morbid obesity BMI > 40
* Untreated chronic GERD
* Pregnancy
* Suspected supraglottic abnormalities
* N2O use
* Need for oral-pharyngeal suctioning
* Undergoing oral and nasal surgery
* Intubation or any oral instrumental manipulations other than
* LMA placements intraoperatively or postoperatively

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Walega, MD, Study Director — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu LQ, Leavitt OS, Malwitz C, Kim H, Doty RA Jr, McCarthy RJ. Comparison of laryngeal mask airway insertion methods, including the external larynx lift with pre-inflated cuff, on postoperative pharyngolaryngeal complications: A randomised clinical trial. Eur J Anaesthesiol. 2017 Jul;34(7):448-455. doi: 10.1097/EJA.0000000000000650. PMID 28590309

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Classic: Group 1 Using the classic inserting technique and completely deflated LMA recommended in the LMA manual.
  Group 1 Classic: Active Comparator: Group 1 classic
  Group 1 Using the classic inserting technique and completely deflated LMA recommended in the LMA manual.
- Group 2 Pre Inflated: Group 2 (pre-inflated): Using the recommended inserting technique with the pre-inflated volume that exists in a LMA from the manufacturer
  Group 2 pre-inflated: Group 2 (pre-inflated): Using the recommended inserting technique with the pre-inflated volume that exists in a LMA from the manufacturer.
Period: Overall Study
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique
Started | 150 | 150 | 150
Completed | 147 | 145 | 149
Not Completed | 3 | 5 | 1
Not completed — Did not receive allocated intervention | 3 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique | Total
Number analyzed (Participants) | 150 | 150 | 150 | 450
Age, Categorical [Count of Participants; unit: Participants] — Population: Some subjects were dropped from the study lost to follow up or the anesthetic management plan changed during the surgical procedure.
  Participants
    number analyzed (Participants) | 147 | 145 | 149 | 441
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 147 | 145 | 149 | 441
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants age in years. Population: Some subjects were dropped from the study lost to follow up or the anesthetic management plan changed during the surgical procedure.
  years
    number analyzed (Participants) | 147 | 145 | 149 | 441
    (all) | 45 (16) | 47 (16) | 46 (16) | 46 (16)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subject number is different because of dropout, lost to follow up or changed anesthetic care.
  Participants
    number analyzed (Participants) | 147 | 145 | 149 | 441
    Female | 58 | 60 | 67 | 185
    Male | 89 | 85 | 82 | 256
Region of Enrollment [Number; unit: participants] — Population: Some subjects were dropped from the study lost to follow up or the anesthetic management plan changed during the surgical procedure.
  participants
    United States: number analyzed (Participants) | 147 | 145 | 149 | 441
    United States | 147 | 145 | 149 | 450
OMA Insertion attempts [Count of Participants; unit: Participants] — The number of total attempts needed to place the airway device. Population: The (N) analyzed is lower because of drop outs and change in anesthesic method during the case.
  Participants
    1 attempt: number analyzed (Participants) | 147 | 145 | 149 | 441
    1 attempt | 122 | 126 | 136 | 384
    2 attempts: number analyzed (Participants) | 147 | 145 | 149 | 441
    2 attempts | 21 | 16 | 12 | 49
    3 attempts: number analyzed (Participants) | 147 | 145 | 149 | 441
    3 attempts | 3 | 3 | 1 | 7
    4 attempts: number analyzed (Participants) | 147 | 145 | 149 | 441
    4 attempts | 1 | 0 | 0 | 1
OSA insertion time in seconds [Median (Inter-Quartile Range); unit: Seconds] — Time in seconds required by the operator to place the airway device. Population: Subjects were lost to follow up or the anesthetic care changed during the surgical procedure.
  Seconds
    number analyzed (Participants) | 147 | 145 | 149 | 441
    (all) | 54 [49 to 67] | 54 [44 to 65] | 56 [46 to 65] | 55 [45 to 65]
Duration of OMA device [Median (Inter-Quartile Range); unit: minutes] — The duration of time in minutes the OMA device was in the larynx. Population: Subjects were lost to follow up or anesthetic management technique changed.
  minutes
    number analyzed (Participants) | 147 | 145 | 149 | 441
    (all) | 71 [50 to 100] | 65 [54 to 105] | 62 [51 to 105] | 66 [50 to 105]
BMI (kg/m∧2 ) [Median (Standard Deviation); unit: BMI (kg/m∧2 )] — BMI (Body Mass Index) (kg/m∧ 2) of participants. Population: Subjects lost to follow up or required a different anesthetic regimen during the surgical procedure.
  BMI (kg/m∧2 )
    number analyzed (Participants) | 147 | 145 | 149 | 441
    (all) | 27.4 (5.2) | 27.7 (5.8) | 27.8 (5.5) | 27.7 (5.6)
Neck Circumference (cm) [Median (Inter-Quartile Range); unit: centimeters] — Neck circumference in centimeters of participants. Population: Some subjects may be have been lost to followup or there was a change in anesthetic care during the surgical procedure.
  centimeters
    number analyzed (Participants) | 147 | 145 | 149 | 441
    (all) | 38 [34 to 41] | 38 [35 to 41] | 38 [34 to 41] | 38 [34 to 41]
Mallampati Class [Number; unit: participants] — Mallampati score or classification is used to predict the ease of endotracheal intubation. Rated on a score of 1 good to 4 poor. Population: Some participants may have been lost to follow up, dropped out or there was a change in anesthetic technique during the surgical procedure
  participants
    Class I: number analyzed (Participants) | 147 | 145 | 149 | 441
    Class I | 69 | 60 | 64 | 193
    Class II: number analyzed (Participants) | 147 | 145 | 149 | 441
    Class II | 39 | 52 | 49 | 140
    Class III: number analyzed (Participants) | 147 | 145 | 149 | 441
    Class III | 20 | 20 | 24 | 64
    Class IV: number analyzed (Participants) | 147 | 145 | 149 | 441
    Class IV | 19 | 13 | 12 | 44
ASA physical status [Number; unit: ASA STATUS] — The ASA physical status classification system is a system for assessing the fitness of a patient prior to a surgical procedure. They include: 1-healthy person.,2-mild systemic disease,3-severe systemic disease,4-severe systemic disease that is a constant threat to life,5- a moribund person who is not expected to survive without the operation and 6- a declared brain-dead person whose organs are being removed for donor purposes. Population: Subject lost to follow up, drop out or there was a change in the anesthetic technique during the surgical procedure.
  ASA STATUS
    ASA l: number analyzed (Participants) | 147 | 145 | 149 | 441
    ASA l | 74 | 70 | 70 | 214
    ASA ll: number analyzed (Participants) | 147 | 145 | 149 | 441
    ASA ll | 67 | 69 | 76 | 212
    ASA lll: number analyzed (Participants) | 147 | 145 | 149 | 441
    ASA lll | 4 | 4 | 3 | 11
    Not documented: number analyzed (Participants) | 147 | 145 | 149 | 441
    Not documented | 2 | 2 | 0 | 4
Surgical Procedure Performed [Number; unit: participants] — Population: Some subjects dropped out. Some of the planned anesthetic techniques were changed during the surgical procedure.
  participants
    Knee Arthroscopy: number analyzed (Participants) | 147 | 145 | 149 | 441
    Knee Arthroscopy | 95 | 85 | 93 | 273
    Shoulder Arthroscopy: number analyzed (Participants) | 147 | 145 | 149 | 441
    Shoulder Arthroscopy | 29 | 42 | 41 | 112
    Elbow Artrhroscopy: number analyzed (Participants) | 147 | 145 | 149 | 441
    Elbow Artrhroscopy | 8 | 6 | 5 | 19
    Other Arthroscopy: number analyzed (Participants) | 147 | 145 | 149 | 441
    Other Arthroscopy | 7 | 3 | 1 | 11
    Breast and skin: number analyzed (Participants) | 147 | 145 | 149 | 441
    Breast and skin | 2 | 4 | 4 | 10
    Hernia Repair: number analyzed (Participants) | 147 | 145 | 149 | 441
    Hernia Repair | 3 | 1 | 3 | 7
    Procedure of the eye: number analyzed (Participants) | 147 | 145 | 149 | 441
    Procedure of the eye | 3 | 3 | 2 | 8
    Other: number analyzed (Participants) | 147 | 145 | 149 | 441
    Other | 0 | 1 | 0 | 1
Perioperative opioid use [Median (Inter-Quartile Range); unit: morphine equivalents milligrams] — Population: Some subjects dropped out. Some anesthetic techniques were changed during the surgical procedure.
  morphine equivalents milligrams
    Intraoperative opioid (morEq milligrams): number analyzed (Participants) | 147 | 145 | 149 | 441
    Intraoperative opioid (morEq milligrams) | 10 [8 to 15] | 10 [6 to 15] | 10 [5 to 15] | 10 [5 to 15]
    Postoperative opioid (morEq milligrams)): number analyzed (Participants) | 147 | 145 | 149 | 441
    Postoperative opioid (morEq milligrams)) | 2.7 [0 to 6.7] | 1.3 [0 to 3.8] | 1.4 [0 to 5] | 1.4 [0 to 6.7]
    Total opioid (morEq milligrams): number analyzed (Participants) | 147 | 145 | 149 | 441
    Total opioid (morEq milligrams) | 15 [10 to 21] | 13 [8 to 18] | 13 [7 to 20] | 13 [7 to 21]
Time to discharge [Median (Inter-Quartile Range); unit: minutes] — Time to discharge is the time admitted into the recovery phase 1 and discharged from the hospital. Population: Some subjects were dropped from the study lost to follow up or the anesthetic management plan changed during the surgical procedure.
  minutes
    Phase 1 immediate PACU (minutes): number analyzed (Participants) | 147 | 145 | 149 | 441
    Phase 1 immediate PACU (minutes) | 67 [54 to 82] | 63 [53 to 79] | 60 [50 to 70] | 63 [50 to 82]
    Phase 2 PACU transition home (minutes): number analyzed (Participants) | 147 | 145 | 149 | 441
    Phase 2 PACU transition home (minutes) | 90 [70 to 120] | 95 [70 to 117] | 95 [65 to 118] | 93 [65 to 120]
    Time to discharge (minutes): number analyzed (Participants) | 147 | 145 | 149 | 441
    Time to discharge (minutes) | 240 [200 to 295] | 236 [193 to 281] | 221 [185 to 283] | 233 [185 to 296]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Present With Postoperative Sore Throat
Description: The primary outcomes for this study will be postoperative pharyngolaryngeal complications of sore throat as reported by the participant.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique
Number analyzed (Participants) | 147 | 145 | 149
Participants | 71 | 71 | 67

2. Primary Outcome: The Primary Outcomes for This Study Will be Postoperative Pharyngolaryngeal Complications Including Dysphonia
Description: The primary outcomes for this study will be postoperative pharyngolaryngeal complications including dysphonia. Difficulty in speaking as assessed by the study team and reported by the participant 24 hours after LMA airway placement.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique
Number analyzed (Participants) | 147 | 145 | 149
Participants | 39 | 31 | 25

3. Primary Outcome: The Primary Outcomes for This Study Will be Postoperative Dysphagia.
Description: The primary outcomes for this study will be postoperative pharyngolaryngeal complication of dysphagia 24 hours after airway placement. This is assessed by a study team member during the 24 hour follow up or reported by the participant.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique
Number analyzed (Participants) | 147 | 145 | 149
Participants | 45 | 38 | 34

4. Primary Outcome: The Primary Outcomes for This Study Will be Postoperative Pharyngolaryngeal Complications Including Dysphagia, Sore Throat and Dysphonia.
Description: The primary outcomes for this study will be postoperative pharyngolaryngeal complications including dysphagia, sore throat and dysphonia 24 hours after airway placement.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique
Number analyzed (Participants) | 147 | 145 | 149
Participants | 83 | 80 | 78
Statistical Analysis 1: Comparison: Group 1 Classic vs Group 2 Pre Inflated vs Group 3 ELL-PIC Technique; We planned a sample size of 429 to achieve a 80% power to detect an effect size difference of w=0.15 using 2 degrees of freedom chi-square test with a significance level (alpha) of .05; Test type: Superiority or Other; p = .76, Chi-squared

5. Secondary Outcome: Severity of Sore Throat
Description: Severity of sore throat 24 hours after airway placement on a 11 point scale of 0-10 ( 0 equals no pain and 10 equals worst pain ever) per recovery hour.
  Low pain = 0 high pain= 500 composite score (0 to 11 points per hour x 24 hours)
Time Frame: 24 hours
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique
Number analyzed (Participants) | 147 | 145 | 149
units on a scale | 143 [30 to 440] | 143 [24 to 440] | 102 [34 to 275]

6. Secondary Outcome: Blood on LMA After Removal
Description: Presence of blood immediately after the removal of the LMA after surgery.
Time Frame: Immediately after LMA removal
Measure: Count of Participants; unit: Participants
Groups:
- Group 3 ELL-PIC Technique: Group 3 (ELL-PIC): Using the ELL-PIC technique.
  Group 3 ELL-PIC Group 3 (ELL-PIC): Using the ELL-PICtechnique
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELL-PIC Technique
Number analyzed (Participants) | 147 | 145 | 149
Participants | 26 | 24 | 13
Statistical Analysis 1: Comparison: Group 1 Classic vs Group 2 Pre Inflated vs Group 3 ELL-PIC Technique; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = .05, Chi-squared; Mean Difference (Final Values) = .02 — The reported p value was calculated

ADVERSE EVENTS:
Time Frame: 24 hours after the airway device removal
Groups:
- Group 3 ELLIA Technique: Group 3 (ELLIA): Using the ELLIA technique.
  Group 3 ELLIA: Group 3 (ELLIA): Using the ELLIA technique
Arm/Group | Group 1 Classic | Group 2 Pre Inflated | Group 3 ELLIA Technique
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/145 | 0/149
Other Adverse Events (participants affected / at risk) | 83/147 | 80/145 | 78/149
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Classic (N=147) | Group 2 Pre Inflated (N=145) | Group 3 ELLIA Technique (N=149)
Postoperative Pharyngolaryngeal Complications Including Dysphagia, Sore Throat and Dysphonia. (Respiratory, thoracic and mediastinal disorders) | 83 (83) | 80 (80) | 78 (78) — Postoperative pharyngolaryngeal complications including dysphagia, sore throat and dysphonia during the timeframe from removal of the airway to 24 hours after the airway removal.
Blood on OMA after removal of the OMA (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 24 (24) | 13 (13) — The presence of blood on the OMA after removal from the airway/

LIMITATIONS AND CAVEATS:
We did not limit the intracuff pressure of the device, but rather used the manufactures recommended volume in the cuff. . There are no current standard of care guidelines for the ideal intracuff pressures within the oropharngolaryngeal mask airway.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No